CLINICAL TRIAL: NCT05796869
Title: The Effect of Laughter Therapy On The Food Craving in Young Women With Premenstrual Syndrome
Brief Title: The Effect of Laughter Therapy On The Food Craving
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinop University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: sınopUmeryem-1
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: PMS; LAUGHTER; Food Habits
Keywords: PMS; Laughter Therapy; Young women; Food Craving
MeSH Terms: conditions — Laughter; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): At the beginning of the study, data collection tools Personal Information Form, Premenstrual Syndrome Scale and Food Craving Scale will be applied to the control group.
  No intervention will be made in the control group. Measurement tools will be applied for the post-test.
- Experimental Group (Experimental): All young women with a Premenstrual Syndrome Scale total score of 110 and above will be included in the study. Since all women who have a Premenstrual Syndrome Diagnostic Scale of 110 and above, volunteer to participate in the study and meet the inclusion criteria will be included in the study, no additional sample selection will be made. The application and control group will be determined on random.org among the group that constitutes the sample of the study. Laughter therapy sessions will be administered face to face to the application group once a week for 2 months by a researcher with a laughter therapy certificate. At the end of two months, the Personal Information Form, Premenstrual Syndrome Scale, and the Food Craving Scale will be administered again to both the application group and the control group.
  Interventions: Behavioral: Assigned Interventions

INTERVENTIONS:
Behavioral: Assigned Interventions — The laughter therapy session will be administered to the application group face to face for 25-30 minutes once a week for 2 months by a researcher with a laughter therapy certificate. In the laughter therapy session, introducing the practitioner and introducing the therapy, breathing exercises for a healthy life, maintaining the rhythm with music, turning laughter that starts like a child's play into reality and meditation practices will be carried out.
  Arms: Experimental Group

SUMMARY:
Premenstrual syndrome (PMS) is characterized by physical, emotional, and behavioral symptoms in the luteal phase that significantly disrupt women's daily lives, including work and personal activities, and resolve spontaneously within a few days of the onset of menstruation. The premenstrual syndrome causes emotional eating, excessive consumption of certain foods, and increased appetite. These unhealthy eating patterns in eating behavior affect health negatively. Women with PMS have an increased appetite and food cravings. It has been stated that the increase in appetite and food cravings are reduced by laughter therapy. Thus, the laughter therapy method, which has no side effects in PMS and negative eating behaviors, can be used and recommended or applied by health professionals.

DETAILED DESCRIPTION:
The universe of the research will be all young women with PMS who study at the designated Faculty of Health Sciences in the Spring semester of the 2022-2023 academic year. The sample of the study will be all young women studying at the Faculty of Health Sciences, meeting the inclusion criteria and agreeing to participate in the study. All young women with a Premenstrual Syndrome Scale total score of 110 and above will be included in the study. Since all women who have a Premenstrual Syndrome Diagnostic Scale of 110 and above, volunteer to participate in the study, and meet the inclusion criteria will be included in the study, no additional sample selection will be made. The application and control group will be determined on random.org among the group that constitutes the sample of the study. Laughter therapy sessions will be applied online for 25-30 minutes once a week for 2 months by the researcher who has the Laughter therapy certificate to the application group. At the end of two months, the Personal Information Form, Premenstrual Syndrome Scale, and the Food Craving Scale will be administered again to both the application group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being a nursing student,
* Being a female student,
* Volunteering to participate in the study.
* Having a PMS score of 43 and above

Exclusion Criteria:

* Not to study as a nursing student
* Being a male student
* Not to volunteer to participate in the study
* Participants who have a PMS score of 42 and below

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Having a PMS score of 43 and above
Enrollment: 90 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Premenstrual Syndrom Scale | One day
  It is a scale developed by Gençdoğan in 2006, measuring the severity of premenstrual symptoms, with a five-point Likert type, containing 44 items and consisting of nine subscales: Depressive Affectiveness, Anxiety, Fatigue, Nervousness, Depressive Thoughts, Pain, Appetite Changes, Sleep Changes and Bloating. When scoring on the scale, "Always" is scored as 5 points, "Often" as 4 points, "Sometimes" as 3 points, "Very little" as 2 points and "Never" as 1 point, and it is evaluated over the total score. The application of the scale is done by retrospectively evaluating the person's "being in the week before menstrual bleeding" situation. The lowest score from the scale is 44 and the highest score is 220. The higher the score, the more severe PMS symptoms are considered. If the person exceeds 50% (110) of the total scale score (220) on the PMS scale, PMS is considered to be present. In the reliability study of the scale, Cronbach's Alpha value was found to be 0.75.

SECONDARY OUTCOMES:
Food Craving: | One day
  The scale was developed by Cepeda-Benito et al. (2000) Akkurt et al. (2019) Turkish validity and reliability were performed. The scale consists of 39 items and is evaluated in a 6-point Likert type. The scale has 9 sub-dimensions. Sub-dimensions and items in sub-dimensions are as follows. "Having Intentions and Plans to Consume Food", "Anticipation of Positive Reinforcement Feelings As a Result of Eating", "Lack of Eating Control Over Eating", "Thoughts or Preoccupation with Food Cravings or Eating", "Craving as a Physiological State", "Emotions That May Be Experienced Before or During Meal", "Cues That May Trigger Food Craving", "Guilt From Cravings and/or for Giving Into Them". The score of each sub-dimension and scale is obtained by dividing the total item scores by the number of items. The scores obtained in this way express the high desire to eat in the scale and in the sub-dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Erdoğan, PhD, Principal Investigator — Sinop University
Locations (1):
- Sinop University, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No